CLINICAL TRIAL: NCT01462643
Title: A 22 Day Controlled, Randomized Clinical Study (PPT) Investigating the Anti-psoriatic Efficacy and the Tolerability of an Ointment Containing a Retinoid and a Steroid in Different Concentrations
Brief Title: Efficacy and Tolerability of LAS41004 Formulations in a Non-occlusive Psoriasis Plaque Test
Acronym: PPT4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Collaborators: proDERM GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H553000-1101; 2011-001384-45 (EudraCT Number)
Record Dates: First submitted 2011-10-04; First posted 2011-10-31 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-10

CONDITIONS: Psoriasis
Keywords: Psoriasis Plaque Test; topical; ointment
MeSH Terms: conditions — Psoriasis | interventions — Steroids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- variant1 (Experimental): topical ointment, once daily application
  Interventions: Drug: LAS41004
- variant 2 (Experimental): topical ointment, once daily application
  Interventions: Drug: LAS41004
- variant 3 (Experimental): topical ointment, once daily application
  Interventions: Drug: LAS41004
- variant4 (Experimental): topical ointment, once daily application
  Interventions: Drug: LAS41004
- variant 5 (Experimental): topical ointment, once daily application
  Interventions: Drug: LAS41004
- variant 6 (Placebo Comparator): topical ointment, once daily application
  Interventions: Drug: LAS41004
- control positive (Active Comparator): topical ointment,once daily application
  Interventions: Drug: LAS41004

INTERVENTIONS:
Drug: LAS41004 — once daily, topical ointment, 100 microgram per day
  Other Names: fixed combinations of retinoid and steroid

SUMMARY:
The aim of the exploratory study is to compare dose related effects of LAS41004 formulations in a non-occlusive PPT.

DETAILED DESCRIPTION:
Going for a non-occlusive application design will allow to draw practical conclusions as being similar to a real treatment situation (compared with a occluded design to maximise effects)

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age
* Caucasian men and women
* Suffering from mild to moderate plaque psoriasis of at least 6 months duration that is amenable to local therapy
* With at least one stable psoriatic plaque in an area sufficient for product application meeting the following criteria:

  1. located at trunk and/or extremities (plaques located on the head, palms, or sole of feet, intertriginous or genitoanal areas are not suitable)
  2. Where more than one plaque is to be used, plaques that are comparable, with at least "2" in each score for scaling, erythema and induration.
  3. No more than 3 points difference in total score (sum of scores for scaling, erythema and induration)
  4. Negative urine pregnancy test (in female patients of child bearing potential)
* In the case of women of childbearing potential, using reliable methods of contraception which result in a low failure rate i.e. less than 1% per year (eg contraceptive implants or injectables, combined oral contraceptives, some intrauterine devices, sexual abstinence or vasectomized partner)

Exclusion Criteria:

* Patients who need systemic treatment for their psoriasis
* Severe forms of psoriasis or forms of psoriasis other than chronic plaque psoriasis, including:
* guttate
* erythroderma
* exfoliative or
* pustular psoriasis
* psoriatic arthritis
* Changes in the expression of psoriasis within the last 6 weeks prior screening
* Intensive UV light exposure within two weeks before the beginning of the test as well as during the study and four weeks after the end of the study at the test area
* Systemic treatment (see table below):

Corticosteroids, antibiotics 4 weeks prior to study day 1 and during conduct of study Retinoids Ciclosporin Methotrexate Fumaric acid esters 3 months prior to study day 1 and during conduct of study Anti-inflammatory substances, NSAIDs 2 weeks prior to study day 1 and during conduct of study Biologics 6 months prior to study day 1 and during conduct of study Planned initiation of, or changes to concomitant medication that could affect Psoriasis (e.g. beta blockers, anti-malaria drugs, lithium) 8 weeks before study start and during study

* Topical treatment of all other body regions with corticosteroids or immunosuppressants where more than 20 % of the body surface area is treated
* Treatment with any non-marketed drug substance within 4 weeks prior to study day 1
* Topical treatment of the test area without adequate time for washout
* Diseases:

Skin infections caused by bacteria, viruses or fungi, including but not limited to tuberculosis, syphilis or varicella zoster infection Parasitic infections Rosacea, perioral dermatitis in test area Moderate or severe illness within the last two weeks before first exposure Other known infectious diseases (e.g. hepatitis or AIDS) Other skin diseases that may confound the evaluation of psoriasis

* Known hypersensitivity to any ingredients of the study drugs,
* Known calcium metabolism disorders
* History of malignancy of any organ system
* Severe impairment of liver or kidney function
* Pregnancy or lactation
* Participation in a clinical trial within the last 30 days prior to the start of this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Decrease of skin thickness(AUC, area under the curve) | day 1 to day 22
  Measurement of skin thickness will be performed by ultrasound (distance between lower border of entry echo and lower border of dermis). The area under the curve, AUC, from day 1 to day 22 will be compared to the reference formulations.

SECONDARY OUTCOMES:
Decrease in scaling | baseline vs day 22
  scoring of scaling (score 0-4) will be performed by investigator
decrease in erythema | baseline vs day 22
  scoring of erythema (score 0-4) wil be performed by investigator
decrease of induration | baseline vs day 22
  scoring of induration (score 0-4) will be performed by investigator
assessment of (s)AE | from baseline to day 22
  a daily record will be performed and if needed the severity and causality assessed

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Willers, MD, Study Director — Almirall Hermal
Locations (1):
- Investigational site, Schenefeld, Germany